CLINICAL TRIAL: NCT07346118
Title: Fluid Balance Guided by Modified Venous Excess Ultrasonography Versus Standard Care in Patients With Acute Kidney Injury Receiving Continuous Renal Replacement Therapy: A Multicentre Randomised Controlled Trial
Brief Title: Fluid Balance Guided by Modified Venous Excess Ultrasonography Versus Standard Care in Patients With Acute Kidney Injury Receiving Continuous Renal Replacement Therapy
Acronym: mVExUS-CRRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0449/2568
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: AKI - Acute Kidney Injury; Fluid Balance; Acute Circulatory Failure; Continuous Renal Replacement Therapy (CRRT); VExUS; Passive Leg Raising; Biomarkers / Blood
Keywords: Acute kidney injury; Fluid balance; Acute circulatory failure; Continuous kidney replacement therapy; mVExUS; Modified Venous Excess Ultrasound; Passive leg raising; Biomarker
MeSH Terms: conditions — Acute Kidney Injury; Shock

STUDY DESIGN:
Intervention Model Description: This will be a multicentre open-label, randomised, controlled trial with parallel groups and balanced computerized randomisation with a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mVExUS-guided fluid management (Active Comparator)
  Interventions: Procedure: mVExUS-guided fluid management
- Standard care (No Intervention)

INTERVENTIONS:
Procedure: mVExUS-guided fluid management — In the intervention arm, mVExUS has to be performed every 24 hours until 72 hours after enrollment. Participants with profile A will have UFNET 0 mL/hr with target fluid balance 0 to +500 mL/day. Patients with profile B will have UFNET 0-20 mL/hr with target fluid balance 0 to -500 mL/day. Patients with profile C will have UFNET 20-40 mL/hr with target fluid balance -500 to -1000 mL/day. Patients with profile D will have UFNET 40-100 mL/hr with target fluid balance neg >1000 mL/day.
  This intervention will be combined with serial lactate monitoring in which lactate levels will be measured every 8 h. When the lactate level rises more than 2 or if there is presence of HIRRT (tachycardia, hypotension, mottling or drop in cardiac index), passing leg raising or mini-fluid challenge (crystalloid fluid bolus 200 mL) will be performed to assess fluid responsiveness. If there is fluid responsiveness, UFNET will be stopped. Once lactate is normalized or episode of HIRRT resolved, the UFNET strat
  Arms: mVExUS-guided fluid management

SUMMARY:
The goal of this randomised controlled trial is to compare the cumulative fluid balance over the first 72 h following inclusion guided by mVExUS versus standard of care in critically ill patients with acute kidney injury receiving CRKT . It will also compare the proportion of CRRT-related complications-including intradialytic hypotension and arrhythmias-between patients managed with mVExUS-guided fluid management and those receiving standard care.

The main questions it aims to answer are:

Does fluid removal rate guided by mVExUS will reduce cumulative fluid balance over the course of the first 72 h of CRRT in ICU patients compared to standard care

Participants will:

Get fluid assessment by mVExUS protocol or a strandard care every 8 hours for 72 hours

DETAILED DESCRIPTION:
After enrollment, the participants have to be randomized within 1 h. In the intervention arm, mVExUS has to be performed every 24 hours until 72 hours after enrollment. Participants with profile A will have UFNET 0 mL/hr with target fluid balance 0 to +500 mL/day. Patients with profile B will have UFNET 0-20 mL/hr with target fluid balance 0 to -500 mL/day. Patients with profile C will have UFNET 20-40 mL/hr with target fluid balance -500 to -1000 mL/day. Patients with profile D will have UFNET 40-100 mL/hr with target fluid balance neg >1000 mL/day.

This intervention will be combined with serial lactate monitoring in which lactate levels will be measured every 8 h. When the lactate level rises more than 2 or if there is presence of HIRRT (tachycardia, hypotension, mottling or drop in cardiac index), passing leg raising or mini-fluid challenge (crystalloid fluid bolus 200 mL) will be performed to assess fluid responsiveness. If there is fluid responsiveness, UFNET will be stopped. Once lactate is normalized or episode of HIRRT resolved, the UFNET strategy has to be restored.

The CRRT technique (haemodialysis, haemofiltration, haemodiafiltration) will be left at the discretion of the treating team. CRRT dose (i.e. dialysate or reinfusion fluids flow rate) will be prescribed at 25-30 ml/kg/hr according to the KDIGO guideline. CRRT dose and UFNET will be indexed to the patient's body weight, and in patients with a body mass index at 30 kg/m2, to the adjusted body weight (calculated as ideal body weight to which will be added 40% of the difference between the actual body weight and the ideal body weight - Du Bois formula). Choice of extra-corporeal circuit anticoagulation (heparin, citrate or none) and implantation site of CRRT catheters will be left at the discretion of the treating physician.

Vasopressors will be titrated as per unit-based protocols to maintain the mean arterial pressure within the bounds prescribed by the physician in charge (most frequently between 65 and 75 mmHg). Indications and category of vasopressors and inotropes will be left at the discretion of the treating team. The diuretic will be stopped once the patient is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years of age)
* Admitted to ICU
* Acute kidney injury by KDIGO criteria
* Initiated CRRT by at least one of the following indications for RRT initiation:
* Serum potassium ≥ 6.0 mmol/L, or
* pH ≤ 7.20 or serum bicarbonate ≤ 12 mmol/L, or
* Evidence of severe respiratory failure, based on a PaO2/FiO2 ≤ 200 and clinical perception of volume overload, or
* Persistent severe AKI (sCr remains > 50% the value recorded at randomization) for > 72 hours from randomization
* Participants giving informed consent

Exclusion Criteria:

* Refuse to participate
* Previous diagnosis of end-stage kidney disease (ESKD) currently on kidney replacement therapy
* Kidney transplant recipient
* Receive RRT before ICU admission within 90 days
* Structural kidney diseases which will interfere with intrarenal doppler ultrasound e.g. renal artery stenosis, autosomal dominant polycystic kidney disease
* Patients with previously known conditions that interfere with portal doppler assessment, namely liver cirrhosis, severe tricuspid regurgitation with structural heart disease or massive ascites.
* Underlying disease process with a life expectancy less than 90 days
* Pregnancy
* Severe cardiac rhythm disturbances (tachyarrhythmia, supraventricular tachycardia)
* Intra-cardiac shunts; Ventricle septal defect, patent foramen ovale, atrial septal defect
* Aortic aneurysm
* Intra-abdominal hypertension (intraabdominal pressure ≥20 mmHg)
* Expected life expectancy <48 hours
* Receiving extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
72-hour cumulative fluid balance between mVExUS-guided management and standard care in critically ill patients with acute kidney injury receiving CRKT. | Hour 0, Hour 72
  In the mVExUS-guided management the fluid removal rate will be guided based on mVExUS ultrasound results. In standard care the fluid removal rate is based on conventionval fluid assessment

SECONDARY OUTCOMES:
28 and 90-day mortality between mVExUS-guided fluid management compared with standard care | 28 days, 90 days
AKI sub-phenotypes, categorized by angiopoietin-1, angiopoietin-2, and soluble TNF receptor-1, association with risk of death in critically ill patients with acute kidney injury receiving CRRT | 28 days
The proportion of CRRT-related complications-including intradialytic hypotension and arrhythmias-between patients managed with mVExUS-guided fluid management and those receiving standard care | Hour 0, Hour 72
The difference patterns of fluid accumulation and net ultrafiltration trajectories and correlation with differences in 28-day mortality in critically ill patients with acute kidney injury receiving CRRT | 28 days

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed will be available from the corresponding author on reasonable request.